CLINICAL TRIAL: NCT05291832
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Explore Perioperative Functional Audio for Anxiety and Cognitive Recovery From Propofol Anaesthesia in Patients Undergoing Endoscopic Procedures
Brief Title: Perioperative Audio for Anaesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brain.fm, Inc. (Industry)
Collaborators: Envision Healthcare (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 001
Record Dates: First submitted 2022-03-14; First posted 2022-03-23 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Anesthesia
Keywords: Music; Anxiety; Recovery
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Conditions are randomly assigned by computer and coded ('A' vs 'B'), where the condition identity is unknown until after data analysis is complete
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brain.fm Music (Experimental): Music with rhythmic amplitude modulation designed to drive neural oscillations.
  Interventions: Other: Brain.fm Music
- Spectrally-matched Noise (Active Comparator): Noise shaped to have the same frequency spectrum (i.e., input level across the cochlea) as the Music condition.
  Interventions: Other: Spectrally-matched Noise

INTERVENTIONS:
Other: Brain.fm Music — Experimental arm
  Arms: Brain.fm Music
Other: Spectrally-matched Noise — Active control arm
  Arms: Spectrally-matched Noise

SUMMARY:
Induction and emergence from propofol can be a difficult process for patients and healthcare workers, and long recovery times in particular can limit the rate of care. A double-blinded randomized controlled trial with 220 patients undergoing elective colonoscopy or endoscopy is proposed to test the impact of perioperative music on patient experience and recovery from propofol anaesthesia. Patients will be assigned at random to hear either rhythmic auditory stimulation (music designed to drive neural oscillations) or spectrally-matched noise (sound that produces the same levels of activity at the cochlea but not expected to drive neural entrainment). Bone-conduction headphones will be administered in pre-operation waiting and will play music (or matched noise) until propofol administration ceases, at which time the music (or noise) will be switched: Pre- and post-operational music is designed to be sedative and stimulative, respectively, created with methods that drive auditory entrainment to promote those states. Outcome measures will be recovery time and the patient's subjective experience (taken via survey).

DETAILED DESCRIPTION:
INTRODUCTION

Can perioperative music improve the patient experience, and speed recovery from propofol anaesthesia?

Difficulties around induction and emergence from general anesthesia are a burden on healthcare workers, and central to a patient's experience. Anxiety prior to a procedure, and confusion upon regaining consciousness, are common experiences that negatively affect both patients and staff. Presurgical anxiety can result in difficulty with intubation and longer presurgical delay periods, burdening nurses and slowing the pace of care. Postsurgically, the duration and quality of a patient's recovery from anesthesia affects healthcare providers and patients, both of whom want to minimize the time spent in the recovery room. Lengthy recovery periods may involve amnesic episodes, delirium, agitation, cognitive dysfunction or other emergence phenomenon, which place strain on patients and staff. Longer recoveries also place strain on the patient's caretaker (e.g., relatives waiting to take them home) and burden the healthcare facility, which may be limited in how quickly procedures can occur based on space available in the recovery area.

Perioperative music has been used effectively to control anxiety and pain (Bringman et al. 2009, Gooding et al. 2012, Tan et al. 2012, Fu et al. 2019,. 2020, 2021), but in these studies the music is chosen to be either relaxing or familiar, with no regard for how it drives brain activity. Prior work has focused on the pre-operative period, and has not considered how stimulative music might be used to kickstart cognition following emergence from anaesthesia. Binaural beats (a type of sound therapy that drives neural entrainment) has been recommended for perioperative use (Padmanabhan et al. 2012), but for relaxation only rather than stimulation. Indeed, no work has been done to distinguish music for induction and emergence, or to provide stimulative music to aid recovery from the unconscious state.

Sound is a powerful neuromodulator, and the auditory system can be used to drive neural activity conducive to a variety of mental states. Part of this effect may be due to how sound (and some music in particular) affects neural oscillations (Will & Berg 2007, Large 2010, Tierney et al. 2014), arousal systems (Thompson et al. 2001, Dillman et al. 2007, Gingras et al. 2014) and dopamine levels (Suttoo et al. 2004, Moraes et al. 2018). Propofol recovery is known to be accelerated by activating the brain's arousal systems via drugs (Chemali et al. 2012) or direct electrical stimulation (Bastos et al. 2021), and music targeting arousal is used to improve cognitive function in humans (Gupta et al. 2018, Woods et al. 2021). Auditory stimulation developed specifically to drive the brain in different ways (Brain.fm music) may be useful perioperatively, and different music may be useful for induction and emergence from anaesthesia.

LITERATURE REVIEW

Propofol recovery Propofol is a widely used general anesthetic agent for ambulatory procedures, but recovery from propofol is not well understood, and the time a patient spends in the recovery room following a procedure may vary widely (Gupta et al. 2004, Shraag et al. 2018). Following return to consciousness (usually characterized by opening the eyes), a patient may experience cognitive deficits or a variety of emergence phenomena such as delirium, aggravation, or amnesia, which are a burden on healthcare workers and likely to be a negative experience for the patient themselves (Lindqvist et al. 2014, Munk et al. 2016, Metterlein et al. 2021). Recovery from propofol can be sped up by activating arousal systems in the brain, for example with methylphenidate (Chemali et al. 2012) or direct thalamic stimulation (Bastos et al. 2021), and by stimuli that have particular arousal value: for example, speaking a patient's name as opposed to other words is more effective at waking patients from propofol, reducing wake-up times by ~20% and reducing time in PACU by ~8% (Jung et al. 2017). Somewhat surprisingly, rather than having negative effects, using arousing stimuli to speed emergence from anaesthesia has been associated with a reduction in emergence delirium in children (Byun et al. 2017). Auditory stimuli like music can also be used to modulate arousal (Husain et al. 2002, Hilz et al. 2014), and sound is commonly used in waking up from sleep. It thus seems likely that stimulating music could be used to speed recovery from general anaesthesia; this point has been noted by others recently but work in this area is still lacking (Seyedalshohadaei et al. 2021).

Perioperative music The role of music in a perioperative setting has largely been confined to anxiety and analgesia, where there is strong evidence for its effectiveness (Bringman et al. 2009, Gooding et al. 2012, Tan et al. 2012, Fu et al. 2019,. 2020, 2021). In a recent example of one such study, Muddanna et al. (2021) tested effects of relaxing music before and during cataract surgery in 165 patients, and found lowered postoperative BP in the test group, along with 48% of the test group reporting feeling 'not at all' or 'a little' anxious (lower ratings of anxiety), versus 30% of the control group. In another study, with 322 patients, Bringman et al. (2009) found that pre-surgical relaxing music was more effective at reducing anxiety than midazlolam (an orally-administered anxiolytic drug). Headsets to reduce anxiety have been tested in clinical settings (Johnson et al. 2012), but use only commercially-available (i.e., not purposely-designed) music, and focus only on relaxation.

Post-operative music has also been found beneficial: in a recent meta-analysis of more than 70 studies, Hole et al. (2015) found strong effects on anxiety, pain, and patient satisfaction, and highly recommended the use of music following surgeries. However, these studies again focus on relaxing music, often of the patient's choice, and in none of these studies was stimulative music used to reduce the duration and difficulty of a patient's emergence from anaesthesia. Studies involving both pre- and post-operative music (Billar et al. 2020, Kappen et al. 2021) use the same music on either side of the procedure, typically with the aim of reducing stress throughout the perioperative period, rather than aiding induction and emergence specifically.

One reason for a lack of interest thus far in stimulative 'wake-up' music may be that music is indeed so effective as an anxiolytic that work in the area has gravitated there. Another possibility is that the use of music to boost arousal or cognition is not widely appreciated, despite having been demonstrated in other contexts such as aiding attentive work (Thompson et al. 2001, Schellenberg et al. 2002, Cassidy et al. 2007), mitigating fatigue (Terry et al. 2020), or improving level-of-consciousness in patients with head trauma (Yekefallah et al. 2021). Finally, the way patients typically return to consciousness in practice may not appear to require external stimulation, since a nurse or doctor will come around to patients at intervals to rouse them (i.e., no 'alarm clock' is needed). However, whether the patient then is able to function cognitively and maintain consciousness (i.e., whether they do in fact wake up when roused), will depend on their neurological state at that time.

Auditory neuromodulation Sound stimuli can modulate brain activity by driving coordinated activity (i.e., entrainment) of neural populations well beyond auditory cortex (Will & Berg 2007, Large 2010, Tierney et al. 2014). This effect is used to drive the brain into states conducive to activities such as sleep (Ngo et al. 2013) or attention (Calderone et al. 2014). Perhaps related to its effect on oscillations, music also can be used to modulate arousal levels bidirectionally (Thompson et al. 2001, Dillman et al. 2007, Gingras et al. 2014). During emergence from propofol, neural oscillations are returning from an altered dynamical state, and changes include increases in beta power (Breshears et al. 2010), an oscillatory band associated with wakefulness and focus (Zanos et al. 2018). Auditory stimuli can be used to shape oscillatory power and may be useful to drive the brain emerging from general anaesthesia. Hunt et al. 2021 used personalized entrainment music (designed to drive oscillations to inhibit pain) on patients with chronic pain, and found a greater improvement than when patients listened to music of their own choosing, demonstrating that the effects of music were due to entrainment rather than affect (emotion or familiarity). Similarly, music designed for sustained attention via entrainment particularly aids listeners with more ADHD-like symptoms (whose oscillatory activity is known to be different), and hightens activity in task-related functional networks (Woods et al. 2021).

In this study we will test music designed to be maximally effective for induction and emergence from propofol (Brain.fm music). The induction (pre-operative) music is designed to induce slow-wave activity and sleep, and has been shown to relax listeners significantly more than commercially-available relaxing music in a pilot study (unpublished). The emergence music (recovery; post-operative) has been shown to drive beta oscillations and improve focus, and as being rated higher in arousal than commercially-available focus music (Woods et al. 2021).

RATIONALE No study to date has explored the possibility of using stimulating music to shorten recovery times from general anaesthesia. One possible reason is that stimulating music is often jarring, which may produce a negative experience for the patient. It may perhaps have been unclear what this music should be, or how it can in practice be delivered during emergence from anaesthesia but not before that point (i.e., stimulating music would be counterproductive during induction). Another reason may be due to practical limitations around placing headphones on the unconscious patient and impacting their situational awareness upon waking. These limitations are overcome in this study, first by having developed a highly-arousing music that drives neural activity strongly, but which is not jarring (i.e., does not have negative emotional valence) by imposing rapid amplitude modulations on music, and secondly by administering this music via bone-conduction headphones which are convenient to place and do not obscure the ear canal. These innovations in content and delivery of music make it possible to test if music can ease a patient's induction and emergence from general anaesthesia, which is a point of concern for both patients and healthcare providers.

The main innovation of this study is to test stimulative music on recovery post-operatively, but we include relaxing music pre-operatively for three reasons: 1) The patient has a reason to apply the headphones themselves (in pre-op waiting), which stay on throughout their procedure. This familiarity with the device might be beneficial for their experience during emergence from anaesthesia. 2) To improve the perioperative experience with a unified music program for the patient; since stimulating music would be counterproductive pre-operatively, relaxing music is used instead. 3) There is some evidence that pre-operative music can reduce the level of anaesthetic agent required during a procedure by reducing anxiety and lowering arousal (LePage et al. 2001, IIkaya et al. 2014; with propofol: Koelsch et al. 2011). Such effects could lead to a faster trajectory of recovery and better patient experience.

The use of relaxing music pre-operatively is thus expected to improve outcome measures, in particular the patient experience more so than recovery times. In the case that the music condition improves patient satisfaction, further studies will be required to explore the contributions of the pre- or post-operative music. However, in the case of improved recovery times, the stimulative music during emergence is more likely to be responsible, and would constitute the first such use of music in a healthcare setting.

RESEARCH QUESTION

Can perioperative music improve the patient experience, and speed recovery from propofol anaesthesia?

OBJECTIVES AND HYPOTHESES

PRIMARY OBJECTIVE AND HYPOTHESIS

Primary Objective:

The primary objective of this study is to explore whether perioperative music-developed to aid induction and emergence from general anaesthesia-can speed recovery times, while maintaining or increasing patient satisfaction with the experience of induction and emergence.

Primary Hypothesis:

If rhythmic auditory stimulation (music developed to drive neural oscillations) improves patient satisfaction with induction and emergence, and speeds recovery from propofol, then these measures should be significantly improved compared to non-rhythmic auditory stimulation (spectrally-matched noise) delivered in the same manner (i.e., through bone-conduction headphones, presented as a recommended aid by a healthcare worker).

STUDY DESIGN

Blind study involving two hundred and twenty (220) participants undergoing elective upper endoscopy or colonoscopy, placed in one of two arms at random. Both groups will receive audio stimulation through bone conduction headphones, starting in the presurgical suite < 2 minutes before application of IV, and ending in the PACU (recovery area) prior to discharge. One group (the test group) will hear Brain.fm music (music designed to be maximally effective for induction and emergence from propofol); the other group (the control group) will hear noise that has been spectrally matched to the Brain.fm music (i.e., contains the same energy at the same frequencies, but is not rhythmic). This control stimulus will be similar to pink noise, which is often used as an auditory stimulus in experiments and is also used by the public to relax and focus. Being spectrally matched to the test music, it will stimulate the cochlea to the same extent and have similar effects in terms of masking (degree of overlap with other sound in the environment).

Bone-conduction headphones will be wireless (bluetooth); audio will be transmitted from an iPad mini attached to the patient's bed (hung from an IV hook; in the clinic only one hook is used for an IV and several are unused); each patient has a given bed from presurgery to recovery. The bone-conduction headphones weigh 26 grams and are low-profile, suitable for lying down (AfterShokz 'Aeropex' model); the iPad mini device size is 5.3" x 7.7".

Staff are required to interact with patients and study equipment with regard to this study at five timepoints:

Headphones applied, audio begins. In the presurgical waiting suite, after the patient has changed into their gown, and just prior to (< 2 minutes) starting the IV. This timing is intended so that the audio will be maximally novel and effective while the IV is being started (a highly anxiety-inducing event for many patients). At this interaction point, the patient is given the bone-conduction device, shown how to wear it, and told it will be on throughout their procedure. They are told they may remove ask to have the device removed by staff at any time if the device or sound is causing discomfort (if they do so, the audio is stopped by staff upon removing the headphones; if this occurs in pre-op their data is excluded from analysis). If they choose to leave it on, they will wake up with it on, and upon waking should leave the device on until they are ready to leave the PACU (unless the device or sound are causing discomfort). They are told that when they take off the device they will be given a very short questionnaire.

Change of audio from sedative to stimulative. After the procedure, propofol is ceased and the attending nurse or anaesthesiologist presses a button on the iPad to switch the audio from sedative to stimulative. After this, the patient is wheeled into PACU.

When wakefulness is noted by staff in PACU, a button is pressed on the iPad. This may be staff confirming wakefulness after an attempt to rouse a patient, or may be staff noticing wakefulness in a patient who has been awake for some seconds or minutes already. As such this measure will not capture the exact wake-up time, but this noise in the data should be hypothesis-independent and non-biasing (i.e., staff will not be more frequently checking on patients with one experimental condition over another; conditions are blinded from the staff).

Headphones removed, audio stopped by staff. After return to consciousness the headphones should stay on until participants are ready to leave the PACU, but the patient may ask to remove them at any time When a patient's headphones are removed (either by request or prior to discharge), the staff will stop the audio, and the three-question survey which appears on the iPad (see Outcome Measures below) will be presented to patients at that point; they are given the option to take it at that pointor any time until they leave the PACU. In the event that a patient asks that their headphones are removed well in advance of leaving the PACU, staff can follow the same procedure, and the data will show that the audio was stopped well before the discharge/headphone-return time. If a patient removes their headphones unsupervised (i.e., staff find a patient with headphones off and do not know how long they have been off), then that patient will be excluded from the dataset.

At the time of discharge (i.e., when the patient leaves their bed), the headphones and iPad are recovered, and a button is pressed on the iPad closing that patient's session. This time is considered the patient's time of discharge.

Randomization between the control and test conditions is implemented by the experiment program on the iPad, which draws a condition at random for each new participant and logs the time of day at each interaction point (the start of audio, switch of audio, wakefulness, headphone removal / playback end, survey completion, and return of equipment). The experiment is double-blinded since the condition a given patient hears is unknown to staff or patient. Since pre-appointment (recruitment) materials do not refer to music but only to auditory stimulation, patients given the noise condition have no indication it is a control condition.

Volume levels are locked to a low, comfortable level, matched across conditions. The bone-conduction device does not obstruct the ear; this in conjunction with a low volume level will ensure patients retain situational awareness and can communicate easily with staff.

The headphones are wiped down with a sterilizing alcohol swab upon being returned to staff, and are placed onto a charging base station. iPads are returned to a charging base station accompanying the headphones. Headphones and iPads are uniquely paired by bluetooth, and so each pair will be labeled (e.g., the headphone set labeled '3' must be used with the iPad labeled '3').

REFERENCES

Bastos, A. M., Donoghue, J. A., Brincat, S. L., Mahnke, M., Yanar, J., Correa, J., ... & Miller, E. K. (2021). Neural effects of propofol-induced unconsciousness and its reversal using thalamic stimulation. Elife, 10, e60824.

Billar, R. J., Kühlmann, A. R., Schnater, J. M., Vlot, J., Tomas, J. J., Zijp, G. W., ... & Wijnen, R. M. (2020). Interventions with Music in PECTus excavatum treatment (IMPECT trial): a study protocol for a randomised controlled trial investigating the clinical effects of perioperative music interventions. BMJ open, 10(7), e036380.

Breshears, J. D., Roland, J. L., Sharma, M., Gaona, C. M., Freudenburg, Z. V., Tempelhoff, R., ... & Leuthardt, E. C. (2010). Stable and dynamic cortical electrophysiology of induction and emergence with propofol anesthesia. Proceedings of the National Academy of Sciences, 107(49), 21170-21175.

Bringman, H., Giesecke, K., Thörne, A., & Bringman, S. (2009). Relaxing music as pre-medication before surgery: a randomised controlled trial. Acta Anaesthesiologica Scandinavica, 53(6), 759-764.

Calderone, D. J., Lakatos, P., Butler, P. D., & Castellanos, F. X. (2014). Entrainment of neural oscillations as a modifiable substrate of attention. Trends in cognitive sciences, 18(6), 300-309.

Cassidy, G., & MacDonald, R. A. (2007). The effect of background music and background noise on the task performance of introverts and extraverts. Psychology of Music, 35(3), 517-537.

Chemali, J. J., Van Dort, C. J., Brown, E. N., & Solt, K. (2012). Active emergence from propofol general anesthesia is induced by methylphenidate. The Journal of the American Society of Anesthesiologists, 116(5), 998-1005.

Dillman Carpentier, F. R., & Potter, R. F. (2007). Effects of music on physiological arousal: Explorations into tempo and genre. Media Psychology, 10(3), 339-363.

Gingras, B., Marin, M. M., & Fitch, W. T. (2014). Beyond intensity: Spectral features effectively predict music-induced subjective arousal. Quarterly Journal of Experimental Psychology, 67(7), 1428-1446.

Gooding, L., Swezey, S., & Zwischenberger, J. B. (2012). Using music interventions in perioperative care. Southern medical journal, 105(9), 486-490.

Gupta, A., Bhushan, B., & Behera, L. (2018). Short-term enhancement of cognitive functions and music: A three-channel model. Scientific reports, 8(1), 1-12.

Gupta, A., Stierer, T., Zuckerman, R., Sakima, N., Parker, S. D., & Fleisher, L. A. (2004). Comparison of recovery profile after ambulatory anesthesia with propofol, isoflurane, sevoflurane and desflurane: a systematic review. Anesthesia & Analgesia, 98(3), 632-641.

Fu, V. X., Oomens, P., Sneiders, D., van den Berg, S. A., Feelders, R. A., Wijnhoven, B. P., & Jeekel, J. (2019). The effect of perioperative music on the stress response to surgery: a meta-analysis. Journal of surgical research, 244, 444-455.

Fu, V. X., Oomens, P., Klimek, M., Verhofstad, M. H., & Jeekel, J. (2020). The effect of perioperative music on medication requirement and hospital length of stay: a meta-analysis. Annals of surgery, 272(6), 961.

Fu, V. X., Sleurink, K. J., Janssen, J. C., Wijnhoven, B. P., Jeekel, J., & Klimek, M. (2021). Perception of auditory stimuli during general anesthesia and its effects on patient outcomes: a systematic review and meta-analysis. Canadian Journal of Anesthesia/Journal canadien d'anesthésie, 1-23.

Henao, D., Navarrete, M., Valderrama, M., & Le Van Quyen, M. (2020). Entrainment and synchronization of brain oscillations to auditory stimulations. Neuroscience research.

Hilz, M. J., Stadler, P., Gryc, T., Nath, J., Habib-Romstoeck, L., Stemper, B., ... & Koehn, J. (2014). Music induces different cardiac autonomic arousal effects in young and older persons. Autonomic Neuroscience, 183, 83-93.

Hole, J., Hirsch, M., Ball, E., & Meads, C. (2015). Music as an aid for postoperative recovery in adults: a systematic review and meta-analysis. The Lancet, 386(10004), 1659-1671.

Hunt, A. M., Fachner, J., Clark-Vetri, R., Raffa, R. B., Rupnow-Kidd, C., Maidhof, C., & Dileo, C. (2021). Neuronal Effects of Listening to Entrainment Music Versus Preferred Music in Patients With Chronic Cancer Pain as Measured via EEG and LORETA Imaging. Frontiers in Psychology, 12, 390.

Husain, G., Thompson, W. F., & Schellenberg, E. G. (2002). Effects of musical tempo and mode on arousal, mood, and spatial abilities. Music perception, 20(2), 151-171.

Ilkkaya, N. K., Ustun, F. E., Sener, E. B., Kaya, C., Ustun, Y. B., Koksal, E., ... & Ozkan, F. (2014). The effects of music, white noise, and ambient noise on sedation and anxiety in patients under spinal anesthesia during surgery. Journal of Perianesthesia Nursing, 29(5), 418-426.

Johnson, B., Raymond, S., & Goss, J. (2012). Perioperative music or headsets to decrease anxiety. Journal of PeriAnesthesia Nursing, 27(3), 146-154.

Jung, Y. S., Paik, H., Min, S. H., Choo, H., Seo, M., Bahk, J. H., & Seo, J. H. (2017). Calling the patient's own name facilitates recovery from general anaesthesia: a randomised double-blind trial. Anaesthesia, 72(2), 197-203.

Kappen, P., Jeekel, J., Dirven, C. M., Klimek, M., Kushner, S., Osse, R. J., ... & Vincent, A. J. (2021). Music to prevent deliriUm during neuroSurgerY (MUSYC) Clinical trial: a study protocol for a randomised controlled trial. BMJ open, 11(10), e048270.

Koelsch, S., Fuermetz, J., Sack, U., Bauer, K., Hohenadel, M., Wiegel, M., ... & Heinke, W. (2011). Effects of music listening on cortisol levels and propofol consumption during spinal anesthesia. Frontiers in psychology, 2, 58.

Large, E. W. (2010). Neurodynamics of music. In Music perception (pp. 201-231). Springer, New York, NY.

Lepage, C., Drolet, P., Girard, M., Grenier, Y., & DeGagné, R. (2001). Music decreases sedative requirements during spinal anesthesia. Anesthesia & Analgesia, 93(4), 912-916.

Lindqvist, M., Schening, A., Granstrom, A., Bjorne, H., & Jakobsson, J. G. (2014). Cognitive recovery after ambulatory anaesthesia based on desflurane or propofol: a prospective randomised study. Acta Anaesthesiologica Scandinavica, 58(9), 1111-1120.

Metterlein, T., Wobbe, T., Brede, E. M., Vogtner, A., Krannich, J., Eichelbrönner, O., & Broscheit, J. (2021). Influencing factors of early cognitive deficits after ambulatory anesthesia. Saudi Journal of Anaesthesia, 15(2), 123.

Moraes, M. M., Rabelo, P. C., Pinto, V. A., Pires, W., Wanner, S. P., Szawka, R. E., & Soares, D. D. (2018). Auditory stimulation by exposure to melodic music increases dopamine and serotonin activities in rat forebrain areas linked to reward and motor control. Neuroscience letters, 673, 73-78.

Munk, L., Andersen, G., & Møller, A. M. (2016). Post-anaesthetic emergence delirium in adults: incidence, predictors and consequences. Acta Anaesthesiologica Scandinavica, 60(8), 1059-1066.

Muddana, S. K., Hess, O. M., Sundar, S., & Venkatesh, R. (2021). Preoperative and perioperative music to reduce anxiety during first-time phacoemulsification cataract surgery in the high-volume setting: randomized controlled trial. Journal of Cataract & Refractive Surgery, 47(4), 471-475.

Nguyen, T., & Grahn, J. A. (2017). Mind your music: The effects of music-induced mood and arousal across different memory tasks. Psychomusicology: Music, Mind, and Brain, 27(2), 81.

Ngo, H. V. V., Martinetz, T., Born, J., & Mölle, M. (2013). Auditory closed-loop stimulation of the sleep slow oscillation enhances memory. Neuron, 78(3), 545-553.

Nilsson, U., Rawal, N., Uneståhl, L. E., Zetterberg, C., & Unosson, M. (2001). Improved recovery after music and therapeutic suggestions during general anaesthesia: a double-blind randomised controlled trial. Acta Anaesthesiologica Scandinavica, 45(7), 812-817.

Padmanabhan, R., Hildreth, A. J., & Laws, D. (2005). A prospective, randomised, controlled study examining binaural beat audio and pre-operative anxiety in patients undergoing general anaesthesia for day case surgery. Anaesthesia, 60(9), 874-877.

Rauscher, F. H., Shaw, G. L., & Ky, K. N. (1993). Music and spatial task performance. Nature, 365(6447), 611-611.

Särkämö, T., Tervaniemi, M., Laitinen, S., Forsblom, A., Soinila, S., Mikkonen, M., ... & Hietanen, M. (2008). Music listening enhances cognitive recovery and mood after middle cerebral artery stroke. Brain, 131(3), 866-876.

Schellenberg, E. G. Music and cognitive abilities. Curr. Dir. Psychol. Sci. 14, 317-320 (2005).

Schraag, S., Pradelli, L., Alsaleh, A. J. O., Bellone, M., Ghetti, G., Chung, T. L., ... & Rehberg, S. (2018). Propofol vs. inhalational agents to maintain general anaesthesia in ambulatory and in-patient surgery: a systematic review and meta-analysis. BMC anesthesiology, 18(1), 1-9.

Seyedalshohadaei, S. M., Baghizadeh, F., & Mirtajani, S. B. (2021) Oblivion Orchestra Hall: How to Facilitate Emergence from Anesthesia with Music. Journal of Cellular & Molecular Anesthesia, 6(3), 279-281.

Shahin, A. J., Trainor, L. J., Roberts, L. E., Backer, K. C., & Miller, L. M. (2010). Development of auditory phase-locked activity for music sounds. Journal of Neurophysiology, 103(1), 218-229.

Suresh, K. P., & Chandrashekara, S. (2012). Sample size estimation and power analysis for clinical research studies. Journal of human reproductive sciences, 5(1), 7.

Sutoo, D. E., & Akiyama, K. (2004). Music improves dopaminergic neurotransmission: demonstration based on the effect of music on blood pressure regulation. Brain research, 1016(2), 255-262.

Tan, D. J. A., Polascik, B. A., Kee, H. M., Hui Lee, A. C., Sultana, R., Kwan, M., ... & Sng, B. L. (2020). The effect of perioperative music listening on patient satisfaction, anxiety, and depression: a Quasi-experimental study. Anesthesiology research and practice, 2020.

Terry, P. C., Karageorghis, C. I., Curran, M. L., Martin, O. V., & Parsons-Smith, R. L. (2020). Effects of music in exercise and sport: A meta-analytic review. Psychological Bulletin, 146(2), 91.

Thompson, W. F., Schellenberg, E. G., & Husain, G. (2001). Arousal, mood, and the Mozart effect. Psychological science, 12(3), 248-251.

Tierney, A., & Kraus, N. (2014). Neural entrainment to the rhythmic structure of music. Journal of Cognitive Neuroscience, 27(2), 400-408.

Will, U., & Berg, E. (2007). Brain wave synchronization and entrainment to periodic acoustic stimuli. Neuroscience letters, 424(1), 55-60.

Woods, K. J., Sempaio, G., James, T., Przysinda, E., Hewett, A., Spencer, A. E., ... & Loui, P. (2021). Stimulating music supports attention in listeners with attentional difficulties. bioRxiv.

Yekefallah, L., Namdar, P., Azimian, J., Mohammadi, S. D., & Mafi, M. (2021). The effects of musical stimulation on the level of consciousness among patients with head trauma hospitalized in intensive care units: A Randomized Control Trial. Complementary Therapies in Clinical Practice, 42, 101258.

Zanos, S., Rembado, I., Chen, D., & Fetz, E. E. (2018). Phase-locked stimulation during cortical beta oscillations produces bidirectional synaptic plasticity in awake monkeys. Current Biology, 28(16), 2515-2526.

ELIGIBILITY:
Inclusion Criteria:

* Opt-in based on recruitment materials.
* English speaking
* Able to consent

Exclusion Criteria:

* Adverse history to anaesthesia
* Cochlear implants
* Hearing aids
* Adverse/unexpected reaction to procedure/anesthesia (post-hoc)
* Headphones accidentally removed during the study period (post-hoc), for example: Data is excluded if playback is stopped before the audio is switched (indicating patient-initiated removal in pre-op); Data is excluded if playback is stopped before wakefulness is noted (indicating accidental removal of headphones)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 329 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2022-07-19 (Actual); Study Completion 2022-07-19 (Actual)

PRIMARY OUTCOMES:
Time to cognitive recovery and discharge | 60 mins
  The time spent in PACU (post-anaesthesia care unit) indicates how quickly patients recovered from propofol anaesthesia. Wakefulness (opening eyes) is noted with a button on the iPad. Audio is to be stopped if headphones are removed. Instead of formal discharge time, nurses are instructed to recover the equipment (iPad) during discharge and end the patient's session (with a button on the iPad). These times logged by the iPad should be coincident with discharge times.
Patient experience | 60 mins
  When either the patient asks to remove the headphones or is ready to leave the PACU, staff retrieve the headphones and press 'stop' on the iPad. This will advance the screen to a three-question survey, which can be completed by the patient at any time between that point and when they leave the PACU. The questions asked are as follows: (1) "I felt anxious immediately before my procedure.", (2) "I feel energized and alert now (following my procedure).", (3) "I would recommend auditory stimulation during this kind of procedure (over one without audio) to friends and family." [Responses as 0-10 horizontal sliders; 0 = Strongly disagree, 5 = Neither Agree nor Disagree, 10 = Strongly Agree]

CONTACTS AND LOCATIONS:
Locations (1):
- Digestive Health Center of Plano, Plano, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided